CLINICAL TRIAL: NCT04992754
Title: Oral Health and Pregnancy : Relation Between Knowledge, Practices and Social Representation of Pregnant Women in the Gynecologie Department at the Montpellier's CHRU
Brief Title: Oral Health and Pregnancy
Acronym: OHAP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0484
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-07

CONDITIONS: Dental Caries; Pregnancy Related
Keywords: Oral hygiene; Public Health; Pregnancy; Prevention; Patients coming to the CHU ADV Montpellier for consultation; Pregnant patients; Knowledge; Literacy
MeSH Terms: conditions — Dental Caries; Literacy | interventions — Psychotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women over 18 years old coming to consult at the gynecology department: Pregnant women over 18 years old coming to consult at the gynecology department in the Montpellier's hospital
  Interventions: Behavioral: psychotherapy, lifestyle counseling

INTERVENTIONS:
Behavioral: psychotherapy, lifestyle counseling — psychotherapy, lifestyle counseling

SUMMARY:
The aim of this study is to identify the knowledge, behavior and social representation on dental health among pregnant women. This study could improve, in the future, prevention, treatments and care for them.

DETAILED DESCRIPTION:
Pregnant women will have to complete a questionnaire that brings together their knowledge, practices and social representations of oral health during their current pregnancy.

ELIGIBILITY:
Inclusion criteria:

* pregnant t women over 18 years old
* French language

Exclusion criteria:

- pregnant women under 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant women over 18 years old in the Montpellier's hospital
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the knowledge | 1 day
  Evaluate the knowledge on the oral health among pregnant woman
Evaluate the practices | 1 day
  Evaluate the practices on the oral health among pregnant woman

SECONDARY OUTCOMES:
Evaluate the social representation | 1 day
  Evaluate the social representation on the oral health among pregnant woman

CONTACTS AND LOCATIONS:
Overall Officials: Camille INQUIMBERT, PhD, Study Director — University Hospital, Montpellier; Camille AMMOR, GRANDATI, resident, Principal Investigator — UH MONTPELLIER
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC